CLINICAL TRIAL: NCT04587102
Title: Whole Body Vibration Training for Diabetic Patients With Burn Injury: RCT
Brief Title: Whole Body Vibration Training for Diabetic Patients With Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ZIZI MOHAMMED IBRAHIM ALI, Assistant Professor of physical therapy, Department of Physical Therapy for Burn and Plastic Surgery, Faculty of Physical Therapy, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIYOBURN
Record Dates: First submitted 2020-08-18; First posted 2020-10-14 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Burn Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: vibration Group (A) will receive low vibrational training in the form of whole body vibration for 8 weeks , while group B is the control, both groups will receive their routine medical care and physical therapy rehabilitation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body viberation :group A (Active Comparator): will receive low vibrational training in the form of whole body vibration for 8 weeks
  Interventions: Other: whole body viberation; Other: Traditional program(balance exercises and resisted exercises)
- control group (B) (Active Comparator): control
  Interventions: Other: Traditional program(balance exercises and resisted exercises)

INTERVENTIONS:
Other: whole body viberation — vibration training in the form of whole body vibration for 20-30 minutes per session, 3 sessions per week for 8 weeks. The vibration training was performed on a whole body vibration platform
  Other Names: WBV
  Arms: whole body viberation :group A
Other: Traditional program(balance exercises and resisted exercises) — balance exercises and resisted exercises

SUMMARY:
Burn injury as well as diabetes mellitus (DM) induce physical functional and psychological impairments. Lower limb burn involving Foot are still a challenging heath condition because of its important sensory role. Balance is disturbed either in patients with lower limb burn injury or diabetic patients. This study aime to compare between the effects whole body vibrational training and Yoga exercises on postural balance, and Activities-specific Balance Confidence in in type II diabetic Patients with foot burn

DETAILED DESCRIPTION:
Thirty eight diabetic patients (17 male, 21female) with foot burn injury, with their age ranged from 40 to 55 years. They will randomly assigned into two equal groups. Group (A) will receive low vibrational training in the form of whole body vibration for 8 weeks (n=19), while group (B) the control group for 8 weeks (n=19) in addition both groups will receive their routine medical care and physical therapy rehabilitation including balancing exercises. Dynamic balance will be evaluated through Biodex balance system (BBS);and balance confidence will be measured by the Activities-specific Balance Confidence Scale (ABC) before the starting and after the end of treatment for all patients in both groups

ELIGIBILITY:
Inclusion Criteria:

* chronic lower limb burns injury for more than 6 months
* Total body surface area (TBSA) burnt ≤ 30%.;

Exclusion Criteria:

* cognitive or mentality dysfunctions,
* psychiatric conditions,
* fractures,
* pregnancy,
* cancer,
* severe vascular complications,
* inability to walk

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Dynamic balance assessment | Change from Baseline at balance scores at 8 weeks
  Biodex Balance System was used to measure the dynamic balance of each patient in both groups (A and B) before and after 8 weeks of treatment.
  The system has a movable balance platform that permits about 20◦ tilt in 360◦ range, and is interfaced with computer software for objective balance assessment. It measures the ability of the patient to control the platform's tilting angle, which is quantified as a variation from the center, as well as the deflection degree over time at different stability levels

SECONDARY OUTCOMES:
The Activities-specific Balance | Change from Baseline at Activities-specific Balance scores at 8 weeks
  A short,six-question version of the Activities-specific Balance scale, the Activities-specific Balance scale. Individuals report their balance confidence in six tasks: standing on tiptoes and reaching for something overhead, standing on a chair to reach for something, being bumped into by people while walking through a mall, stepping off an escalator holding onto the railing, stepping off an escalator without holding onto the railing, and walking on an icy sidewalk ABC scores range between 0% and 100%, with higher scores indicating better balance confidence

CONTACTS AND LOCATIONS:
Overall Officials: ZIZI MOHAMMED I ALI, Principal Investigator — Cairo University
Locations (3):
- Egypt (2):
  - Zizi Mohammed Ibrahim Ali, Giza, Nnjkjk
  - Burn Unit at Om El Masrien Hospital, Giza
- Zizi Mohammed Ibrahim Ali, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No